CLINICAL TRIAL: NCT04001972
Title: Intervention Combining Interactive Communication Technologies and Nicotine Replacement Therapy Sampling for Proactively Recruited Smokers in Smoking Hotspots: a Pragmatic Randomized Controlled Trial
Brief Title: Interactive Communication Technologies and Nicotine Replacement Therapy Sampling for Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICTNRT
Record Dates: First submitted 2019-06-12; First posted 2019-06-28 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Smoking Cessation; Tobacco Use Cessation
Keywords: tobacco dependence treatment; combined brief intervention; AWARD advice; active referral; nicotine replacement therapy; information and communication technologies
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation | interventions — Crisis Intervention; corticosteroid hormone-induced factor; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Brief advice (AWARD model) + NRT-S + IM Apps and Chatbot
  Interventions: Behavioral: Brief advice (AWARD model); Drug: NRT-S; Behavioral: IM Apps and Chatbot
- Control group (Active Comparator): Brief advice (AWARD model) + regular SMS
  Interventions: Behavioral: Brief advice (AWARD model); Behavioral: Regular SMS message

INTERVENTIONS:
Behavioral: Brief advice (AWARD model) — Ask: smoking habit, quit intention and attempt, smoking reduction intention, previous quitting experience including NRT and SC use.
  Warn: smokers will be orally warned about the harms of smoking and receive a A5-sized leaflet, which includes some shocking pictures of smoking-related diseases, and SC services information.
  Advise: smokers will be advised to quit as soon as possible and use NRT or SC services.
  Refer: smokers will be encouraged to seek SC services for free NRT or other SC services. Those who agreed will be actively referred to their preferred SC services. The collected contact information with consent will be sent to the SC services providers for a quick appointment and follow-up.
  Do-it-again: Relapsed smokers (identified during follow-ups and IM conversation) will receive the "Advise" and "Refer" intervention.
  Other Names: Ask, Warn, Advise, Refer and Do-it-again
Drug: NRT-S — One-week free NRT (gum or patch) will be provided with dosage based on time to first cigarette smoking after waking up in the morning and previous NRT use (standard practice and according to specific NRT product instructions). Subjects who have first cigarette <30 minutes in the morning or have previously used NRT, will receive 4mg nicotine gum or 21mg nicotine patch. Those who have first cigarette >30 minutes after waking up and have not previously used NRT will receive 2mg nicotine gum or 14mg nicotine patch. NRT use and potential side effects will be briefly explained orally based on standardized script according to the product instructions. An NRT use card containing reminders of NRT use and potential side effects will be given.
  Other Names: NRT sample
  Arms: Intervention group
Behavioral: IM Apps and Chatbot — Twelve-week personalized behavioral support will be delivered using interactive communication technologies using (1) regular tailored messages on abstinence, and (2) synchronous IM Apps conversation with trained SC advisors, and (3) a Chatbot: A Chatbot will be built using open source NLP and machine intelligence platforms. The unstructured text data from our previous study (ClinicalTrials.gov ID: NCT03182790) will be used to train the proposed Chatbot. We will draft responses for each identified question. The final version will be incorporated with Application Programming Interface (API) integration into user-friendly apps (iOS/Android/web app) with a backend server support and continuous data collection for potential bigdata analysis.
  Arms: Intervention group
Behavioral: Regular SMS message — Regular SMS messages focus on general health and remind the importance of participating in the follow-up surveys and biochemical validation for quitting
  Arms: Control group

SUMMARY:
Brief advice combined with active referral to smoking cessation (SC) services increases quitting. We aim to strengthen the effect of combined intervention by using interactive communication technologies and nicotine replacement therapy sampling (NRT-S).

DETAILED DESCRIPTION:
Objectives: Brief advice combined with active referral to smoking cessation (SC) services increases quitting. We aim to strengthen the effect of combined intervention by using interactive communication technologies and nicotine replacement therapy sampling (NRT-S).

Design and subjects: Pragmatic, individual randomized controlled trial in 664 daily smokers proactively recruited in smoking hotspots in Hong Kong.

Interventions: Subjects in the Intervention group will receive face-to-face brief advice (including SC services referral) using AWARD model and 1-week free NRT sample (NRT-S) at baseline; and 12-week personalized behavioral support using interactive communication technologies (include regular tailored messages on abstinence, and synchronous IM Apps [e.g. WhatsApp] conversation with trained SC advisors and a Chatbot). Subjects in the Control group will receive the same AWARD advice without NRT-S at baseline, and regular short-message-service messages on general health and reminders to participate in follow-up.

Main outcome measures: Primary outcomes are carbon monoxide validated smoking abstinence at 6-month and 12-month. Secondary outcomes include self-reported past 7-day abstinence, smoking reduction, quit attempt, SC services use, NRT use, self-efficacy on quitting and quality of life.

Data analysis: Intention-to-treat and cost-effectiveness analyses will be conducted. Mediation analyses will explore the underlying mechanisms of Chatbot and IM Apps behavioral support to promote quitting. Individual interviews with quitters and non-quitters, and content analysis of Chatbot/IM Apps will be conducted to have in-depth understanding on the effects of intervention on various outcomes.

Expected results: The Intervention group will have statistically significant higher validated smoking abstinence rates than the Control group at 6-month and 12-month.

ELIGIBILITY:
Inclusion Criteria:

1. Adult smokers aged 18+ years who smoke cigarette(s) daily.
2. Exhaled carbon monoxide (CO) level of ≥ 4ppm.
3. Having smartphones and willing to install IM Apps and a Chatbot.
4. Hong Kong residents able to read and communicate in Chinese (Cantonese or Putonghua).

Exclusion Criteria:

1. Smokers who have psychiatric/psychological diseases/on regular psychotropic medications.
2. Smokers who are using SC medication, NRT, other SC services or projects.
3. Smokers who have contraindication for NRT use: severe angina, arrhythmia, myocardia infraction, pregnancy (or intended to become pregnant <6 months) or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Biochemically validated abstinence of NRT-S +IM Apps and Chatbot vs. regular SMS | At 6-month follow-up
  NRT-S +IM Apps and Chatbot vs. regular SMS on validated abstinence defined as exhaled carbon monoxide <4ppm
Biochemically validated abstinence of NRT-S +IM Apps and Chatbot vs. regular SMS | At 12-month follow-up
  NRT-S +IM Apps and Chatbot vs. regular SMS on validated abstinence defined as exhaled carbon monoxide <4ppm

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence abstinence | At 6-month follow-up
  Self-reported no cigarette smoking (even a single puff) in the past 7 days
Self-reported 7-day point prevalence abstinence | At 12-month follow-up
  Self-reported no cigarette smoking (even a single puff) in the past 7 days
Self-reported past 24-week continuous abstinence | At 6-month follow-up
  Self-reported no cigarette smoking (even a single puff) in the past 24 weeks
Self-reported past 24-week continuous abstinence | At 12-month follow-up
  Self-reported no cigarette smoking (even a single puff) in the past 24 weeks
Planned quit day | At 6-month follow-up
  Planned quit day with responses "within 7 days/within 30 days/within 60 days/undecided"
Planned quit day | At 12-month follow-up
  Planned quit day with responses "within 7 days/within 30 days/within 60 days/undecided"
Change in number of quit attempts from baseline | At 6-month follow-up
  Defined by abstinence for at least 24 hours from baseline
Change in number of quit attempts from baseline | At 12-month follow-up
  Defined by abstinence for at least 24 hours from baseline
Change in smoking reduction rate from baseline | At 6-month follow-up
  Defined by at least 50% reduction in baseline daily number of cigarettes
Change in smoking reduction rate from baseline | At 12-month follow-up
  Defined by at least 50% reduction in baseline daily number of cigarettes
Change in micotine addiction level from baseline | At 6-month follow-up
  Assessed by Heaviness of Smoking Index (range 0 to 6 with higher score indicating greater nicotine dependence)
Change in micotine addiction level from baseline | At 12-month follow-up
  Assessed by Heaviness of Smoking Index (range 0 to 6 with higher score indicating greater nicotine dependence)
Any access to a smoking cessation service | At 6-month follow-up
  Any access to a smoking cessation service with responses "yes/no"
Any access to a smoking cessation service | At 12-month follow-up
  Any access to a smoking cessation service with responses "yes/no"
Any use of nicotine replacement therapy | At 6-month follow-up
  Any use of nicotine replacement therapy with responses "yes/no"
Any use of nicotine replacement therapy | At 12-month follow-up
  Any use of nicotine replacement therapy with responses "yes/no"
Change in quality-adjusted life year (QALY) | At 12-month follow-up
  Change in quality-adjusted life year (QALY) will be estimated using the validated Chinese five-level EuroQol five-dimensional questionnaire (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo N, Luk TT, Wu YS, Guo Z, Chu JCL, Cheung YTD, Chan CHH, Kwok TTO, Wong VYL, Wong CKH, Lee JJ, Kwok YK, Viswanath K, Lam TH, Wang MP. Effect of mobile interventions with nicotine replacement therapy sampling on long-term smoking cessation in community smokers: A pragmatic randomized clinical trial. Tob Induc Dis. 2023 Mar 24;21:44. doi: 10.18332/tid/160168. eCollection 2023. PMID 36969982